CLINICAL TRIAL: NCT00448500
Title: Measurement of Biomarkers in the Exhaled Breath Condensate in Patients With Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Brief Title: Exhaled Breath Condensate (EBC) Assessment in Acute Exacerbation of Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Fanny WS Ko, The Chinese University of Hong Kong
Other Study IDs: Resp/ko/2006/004
Record Dates: First submitted 2007-03-14; First posted 2007-03-16 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; exhaled breath condenate; Exhaled breath condenate, acute exacerbation of COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Exhaled breath condensate
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aimed to assess airway inflammation in patients during the course of acute exacerbations of chronic obstructive pulmonary disease (AECOPD) by serial analyses of their exhaled breath condensates (EBC).

DETAILED DESCRIPTION:
Subject recruitment

Patients who had been admitted to the Prince of Wales Hospital with AECOPD were recruited for this study. Subjects with pneumonic changes on the chest radiographs were excluded. Age and sex-matched COPD subjects at stable state (without AECOPD for at least 10 weeks) and healthy, non-smoking subjects were recruited as controls.

Collection of exhaled breath condensate (EBC) EBC was collected using the EcoScreen (VIASYS Healthcare, Conshohochen, PA, USA) according to the manufacturer's instructions. EBC was stored in 250 microL aliquots immediately at -70oC until analysis. EBC was collected on Day 5, 14, 30 and 60 after hospitalization for subjects with AECOPD. For the stable COPD patients and normal controls, EBC collection was performed once.

Measurement of TNF alpha, LTB4 and IL-8 The concentrations of TNF alpha, LTB4, and IL-8 in EBC were measured in one batch by high-sensitivity sandwich enzyme immunoassays (TNF alpha and IL-8 from BioSource International, Camarillo, CA, USA; LTB4 from Cayman Chemical Company, Ann Arbor, MI, USA) according to the manufacturers' instructions. Intra-subject repeatability of TNF alpha, LTB4 and IL-8 was assessed by collection of EBC in stable COPD subjects. EBC was collected as described above at the same time (09:00 to 10:00) on 2 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had been admitted to the Prince of Wales Hospital with AECOPD were recruited for this study. AECOPD was defined when a patient with background COPD according to the GOLD guideline presented with at least two of the following major symptoms (increased dyspnoea, increased sputum purulence, increased sputum volume) or one major and one minor symptom (nasal discharge/congestion, wheeze, sore throat, cough) for at least two consecutive days.
* Age and sex-matched COPD subjects at stable state (without AECOPD for at least 10 weeks) and healthy, non-smoking subjects were recruited as controls. Current smokers (defined as cigarette smoking in the last 6 months) were excluded from this study.

Exclusion Criteria:

* Subjects with pneumonic changes on the chest radiographs were excluded.
* Current smokers (defined as cigarette smoking in the last 6 months) were excluded from this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD patients with exacerbations Stable COPD patients Normal subjects
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2006-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fanny WS Ko, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong